CLINICAL TRIAL: NCT00359073
Title: Effect of Montelukast on Experimentally-Induced RV16 Infection in Volunteers With Mild Asthma
Brief Title: Effect of Montelukast on Experimentally-Induced RV16 Infection in Asthma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: H-2006-0173; 31799 (Other: PI)
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-03

CONDITIONS: Asthma
Keywords: asthma; leukotrienes; rhinovirus
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Montelukast (Active Comparator): montelukast (10 mg everyday)
  Interventions: Drug: montelukast
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: montelukast — 10 mg everyday
  Other Names: Singulair
  Arms: Montelukast
Drug: placebo — like placebo
  Other Names: like placebo
  Arms: Placebo

SUMMARY:
People with asthma may have asthma worsening when they have an upper respiratory infection due to a virus or a common cold. Leukotrienes are increased in nasal secretions from children with Respiratory Syncytial Virus (RSV) and lung washings during times of acute lung inflammation. Experimental virus exposure in adults is also associated with increases in nasal leukotrienes.

The degree to which leukotrienes play a role in asthma worsening is unknown.There is information linking leukotrienes to viral infections, allergic inflammation, and asthma exacerbation.This information supports the hypothesis that virus-induced leukotrienes contribute to the severity of respiratory infections and in susceptible individuals, lead to lower airway obstruction and exacerbations of asthma. We propose to use montelukast in an experimental viral challenge model to explore this hypothesis.

DETAILED DESCRIPTION:
Viral infections are important causes of wheezing illnesses throughout childhood and in adults with asthma. There has been progress in identifying mechanisms and risk factors for severe respiratory symptoms, and in particular, wheezing. Given this close relationship, it would be attractive to apply antiviral strategies to the prevention and treatment of asthma, and both RV and RSV are obvious targets. Unfortunately, attempts at developing an RSV vaccine have so far been unsuccessful, and vaccination to prevent RV infection does not seem to be feasible due to the large number of serotypes. Antiviral medications have been tested in clinical trials, however one problem with this approach is that once the clinical signs and symptoms appear, viral replication is well underway.

The other potential therapeutic approach for respiratory viral infections would be to selectively inhibit pro-inflammatory immune responses induced by the virus. The beneficial effects of systemic glucocorticoids indicate that this approach is valid; the challenge will be to develop treatments with greater efficacy and a reduced potential for adverse effects. The large body of information linking cysteinyl leukotrienes to viral infections, allergic inflammation, and asthma exacerbations, strongly supports the hypothesis that virus-induced leukotrienes contribute to the severity of respiratory infections and in susceptible individuals, lead to lower airway obstruction and exacerbations of asthma. We propose to use montelukast in an experimental viral challenge model to explore this hypothesis.

ELIGIBILITY:
Inclusion Criteria:

A subject with mild persistent asthma is eligible for participation in the study if all of the following inclusion criteria apply:

* Male or female with no health concerns that might affect the outcome of the study
* Age 18-65 range
* diagnosis of mild persistent asthma based on clinical findings such as cough, wheeze and shortness of breath
* a history of asthma for at least six months prior to screening
* FEV1> 80% of predicted
* presence of allergy based on at least one positive prick skin test when tested with a standard panel of common allergens
* ability to produce sputum when induced during the baseline assessments
* asthma medications consisting of only inhaled short acting B-agonist taken as needed
* reversible airways disease as indicated by > 12% reversibility post B-agonist or
* methacholine hyperresponsiveness (PC20 < 8 mg/ml)
* ability to give valid informed consent to participate by signing and dating a written consent form

Exclusion Criteria:

A subject is not eligible to participate in this study if any of the following exclusion criteria apply:

* History of severe episodes of asthma with respiratory infections
* Screening serum RV16 antibody titer > 1
* Current smoker or has a smoking history exceeding 5 pack years
* Currently receiving immunotherapy
* Currently participating in another clinical trial or has participated in an investigational drug trial within one month of screening
* Unable, in the judgment of the investigator, to comply with directions and/or tolerate the procedures required for participation in this trial
* Pregnant or breast-feeding or has a planned pregnancy during the course of the study
* Regular use of an asthma controller such as montelukast or an inhaled corticosteroid.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-10 (Actual); Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James E Gern, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kloepfer KM, DeMore JP, Vrtis RF, Swenson CA, Gaworski KL, Bork JA, Evans MD, Gern JE. Effects of montelukast on patients with asthma after experimental inoculation with human rhinovirus 16. Ann Allergy Asthma Immunol. 2011 Mar;106(3):252-7. doi: 10.1016/j.anai.2010.11.021. Epub 2011 Jan 13. PMID 21354028
- See also: Allergy,Asthma and Pulmonary Clinical Research Unit website — http://www.medicine.wisc.edu/asthma/asthmamain

RESULTS

PARTICIPANT FLOW:
Groups:
- Montelukast: subjects received study drug montelukast, 10 mg once per day
- Placebo: subjects received placebo, once per day
Period: Overall Study
Arm/Group | Montelukast | Placebo
Started | 12 | 13
Completed | 8 | 11
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Eligibility criteria no longer met | 3 | 0
Not completed — developed RV16 antibody | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Montelukast | Placebo | Total
Number analyzed (Participants) | 8 | 11 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 20 (2) | 21 (3) | 20 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 7
  Male | 5 | 7 | 12
Region of Enrollment [Number; unit: participants]
  United States | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Asthma Symptom Score
Description: Asthma symptom scores were assessed twice per day with subjects completing a validated daytime diary card before bed and a nocturnal diary card on awakening. Subjects answered 4 questions about their asthma symptoms (0, none of the time; 6, all of the time). Daily score were calculated as the average of the 4 questions and an overall score for the week was assessed as the average of the daily scores. Time frame measurement was Day 7.
Time Frame: Day 7
Measure: Median (Inter-Quartile Range); unit: Asthma symptom score
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 8 | 11
Asthma symptom score | 2.3 [0.0 to 4.9] | 2.1 [0.1 to 4.1]

2. Secondary Outcome: Peak Viral Shedding
Description: Viral shedding was measured in both groups. Viral titers from nasal lavage were calculated after 4 tissue culture tubes containing WI38 cells (human lung diploid cells) were inoculated for each serial 10-fold dilution of samples and incubated while rolling at 33 degrees Celsius for 10 days (measurement for analysis was taken at baseline and 7 days). Tubes were read at baseline and 7 days later. TCID50 was calculated as the concentration that was capable of infecting 50% of the tubes. Viral titers are expressed as TCID50 per milliliter. Time frame measurement was at baseline and 7 days.
Time Frame: Baseline and 7 days
Measure: Median (Inter-Quartile Range); unit: TCID50 per milliliter
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 8 | 11
TCID50 per milliliter | 2.5 [2.3 to 4.5] | 3.5 [2.5 to 4.5]

3. Secondary Outcome: Sputum Eosinophil Count
Description: Sputum was collected from both groups over 14 days after inoculation with the cold virus. Cell counts and differentials were made from sputum samples after treatment with 0.1% dithiothreitol. Eosinophils were counted and are expressed as as percentage of cells (percent of the total number counted) at the 14 day timepoint.
Time Frame: 14 days
Measure: Median (Inter-Quartile Range); unit: percentage of eosinophils
Arm/Group | Montelukast | Placebo
Number analyzed (Participants) | 8 | 11
percentage of eosinophils | 0.3 [0.1 to 0.3] | 2.0 [0.3 to 2.7]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Montelukast | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/11
Other Adverse Events (participants affected / at risk) | 1/8 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Montelukast (N=8) | Placebo (N=11)
Upper Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (General disorders) | 1 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Was a pilot study; small sample size limited statistical power; subgroup analysis not applicable

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No